CLINICAL TRIAL: NCT06236945
Title: Composite Autonomic Scoring Scale and HUTT to Assess Cardiac Autonomic Nervous Function: A Preliminary Study
Brief Title: HUTT to Assess Cardiac Autonomic Nervous Function
Status: Recruiting | Type: Observational
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Yan Ding, Head of Neurology, The First Hospital of Hebei Medical University
Other Study IDs: 20230213
Record Dates: First submitted 2023-12-27; First posted 2024-02-01 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Autonomic Nervous System Diseases
MeSH Terms: conditions — Autonomic Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Autonomic nervous system diseases can cause abnormalities in the circulatory system, leading to malignant arrhythmia and sudden cardiac death. Standardized, operable, and simplified diagnostic indicators are urgently needed to evaluate autonomic nervous function, particularly cardiac autonomic nervous function. The investigators use HUTT in order to provide data support for cardiac autonomic nervous system evaluation.

DETAILED DESCRIPTION:
In this study, 169 samples with vertical tilt test and 24-h Holter ECG data from February 13, 2023 to October 31, 2023 were selected. The AC, DC, and 24-h HRV were compared with the CASS to identify the indicators with the strongest correlation with the CASS sympathetic and vagus nerve scores. The best index was selected, and the score intervals were delimited. The sensitivity and specificity of the defined vagal and sympathetic intervals were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Vertical tilt test and 24-hour holter electrocardiogram were performed at the same time

  * Receive treatment in our hospital.

Exclusion Criteria:

* Taking benzodiazepines or hypotensive drugs within 24 hours

  * Combined with mental illness, severe dementia, serious organ disease

    * Severe arrhythmia, deep breathing and poor coordination of Valsaval movements affected the interpretation of results.

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 1122 (546 males, 576 females) samples were collected according to the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 1122 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To find the indicators which are most correlated to the sympathetic and vagus nerves. | February 13, 2023 to December 31, 2025
  The investigators use HUTT and CASS score to find some indicators which are most correlated to the sympathetic and vagus nerves,so that can give data support to the clinical treatments

CONTACTS AND LOCATIONS:
Overall Officials: Yan Ding, M.D., Principal Investigator — Department of Neurology，Xuanwu Hospital，Capital Medical University，Beijing，China.
Locations (1):
- The First Hospital Of Hebei Medical University, Shijiazhuang, Hebei, China